CLINICAL TRIAL: NCT01815346
Title: A Phase I-II Study of Acupuncture for the Treatment of Chronic, Taxane-Induced Peripheral Neuropathy in Breast Cancer Survivors
Brief Title: Acupuncture Chemotherapy-Induced Peripheral Neuropathy (CIPN) IRG
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-1054; NCI-2014-01520 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-03-15; First posted 2013-03-21 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Breast cancer survivors; Chronic, taxane-based chemotherapy-induced peripheral neuropathy; CIPN; Acupuncture treatments; Quality of life; Hand function; Balance; Questionnaires; Surveys
MeSH Terms: conditions — Breast Neoplasms; Bronchiolitis Obliterans Syndrome | interventions — Acupuncture Therapy; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture Group - Twice a Week (Experimental): Acupuncture 2 times a week for 6 weeks. Participants receive acupuncture to the arms, legs, and abdomen. The acupuncture needles will be left in place for about 20 minutes.
  Interventions: Procedure: Acupuncture; Behavioral: Questionnaires; Other: Hand Function and Balance Tests
- Acupuncture Group - Three Times a Week (Experimental): Acupuncture 3 times a week for 4 weeks. Participants receive acupuncture to the arms, legs, and abdomen. The acupuncture needles will be left in place for about 20 minutes.
  Interventions: Procedure: Acupuncture; Behavioral: Questionnaires; Other: Hand Function and Balance Tests

INTERVENTIONS:
Procedure: Acupuncture — One group receives acupuncture 2 times a week for 6 weeks.
  One group receives acupuncture 3 times a week for 4 weeks.
  Participants receive acupuncture to the arms, legs, and abdomen. The acupuncture needles will be left in place for about 20 minutes.
Behavioral: Questionnaires — Three questionnaires completed at baseline, midpoint, and four weeks after completion of acupuncture treatment.
  Other Names: Surveys
Other: Hand Function and Balance Tests — Tests completed at baseline, midpoint, and four weeks after completion of acupuncture treatment. These tests should take about 20 minutes to complete.

SUMMARY:
The goal of this clinical research study is to compare the level of effectiveness for 2 acupuncture treatment schedules for chronic CIPN in breast cancer survivors. Researchers also want to study how patients may respond to acupuncture treatments, and how the treatments may affect quality of life, hand function, balance, and the use of drugs for neuropathy pain.

DETAILED DESCRIPTION:
Peripheral neuropathy is one of the most common chemotherapy side effects affecting the nerves. Each year, thousands of patients receive taxane-based chemotherapy and more than 50-60% of these patients will have CIPN. CIPN can cause painful or abnormal skin sensation (such as pins and needles), numbness, and/or nerve damage that may affect movement.

Baseline Visit:

You have already had certain tests as part of your routine care that helped show that you were eligible to take part in this study. If you agree to take part in this study, the following tests and procedures will be performed at your first study visit:

* Your vital signs (blood pressure, heart rate, temperature, and breathing rate) will be measured.
* Your medical history will be recorded.
* You will be asked about any drugs you may be taking and any side effects you may be having.
* You will complete 3 questionnaires about any symptoms you may have. The questionnaires should take about 15-30 minutes to complete in total.
* You will perform hand function and balance tests. For these tests, you will complete tasks such as putting pegs into a pegboard. These tests should take about 20 minutes to complete.

Study Groups:

You will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. Both groups will receive a total of 12 acupuncture treatments.

* Group 1 will receive acupuncture 2 times a week for 6 weeks.
* Group 2 will receive acupuncture 3 times a week for 4 weeks.

Acupuncture Treatments (All Participants):

Your acupuncture treatments will be given on an outpatient basis in private rooms. For the treatment, you will lay down on a table face up. The acupuncturist will disinfect the selected acupuncture points with alcohol. Then, the acupuncture needles will be placed so that you achieve a "de qi" sensation, which is often described as an achy, tingling, or numb feeling of pressure after an acupuncture needle has been properly placed in the skin.

The acupuncture needles will be left in place for about 20 minutes. During this time, the needles will be charged with a small electric current, which is done to enhance the effect of the acupuncture treatment. The needles may also be twirled to cause the sensation of de qi.

During each treatment session, you will receive acupuncture to the arms, legs, and abdomen.

Study Visits:

One (1) time every week:

* Your vital signs will be measured.
* You will be asked about any drugs you may be taking and any side effects you may be having.

At Weeks 3 and 6 (Group 1 only) and Weeks 2 and 4 (Group 2 only):

* You will complete the same 3 questionnaires you completed at baseline.
* You will perform hand function and balance tests.

Length of Study:

You may continue your participation on this study for up to 10 weeks, as long as the study doctor thinks it is your best interest. Your active participation in this study will be over after you have completed the 4-week follow-up visit.

Follow-Up:

Four (4) weeks after you complete the acupuncture treatment, the following tests and/or procedures will be performed:

* Your vital signs will be measured.
* Your medical history will be reviewed and any updates will be recorded.
* You will be asked about any drugs you may be taking and any side effects you may be having.
* You will complete the same 3 questionnaires you completed at baseline.
* You will perform hand function and balance tests.

This is an investigational study. The acupuncture needles being used in this study are FDA approved for medical use. The use of acupuncture treatments for chronic CIPN on the schedules in this study is investigational.

Up to 54 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have the ability to understand English, sign a written informed consent document, and be willing to follow protocol requirements.
2. Age >/= 18 years.
3. History of a diagnosis of breast cancer.
4. Patients must have neuropathy greater or equal to 2 according to CTCAE v 4.0 scale, clinically evaluated within 30 days of consent, despite previous treatment, which may include Neurontin, Cymbalta and/or Lyrica for at least 30 days. Patients receiving any of these drugs must remain on the same medications throughout the study period; however, adjustments in dosage are allowed. Patients are allowed to stop medications but not replace them with other medications.
5. The patient's previous chemotherapy treatment must have included a taxane (paclitaxel, nab-paclitaxel, or docetaxel) and considered the primary cause of the neuropathy by the medical team.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2.
7. Ability to complete the 4 or 6 weeks of acupuncture and follow-up assessments.

Exclusion Criteria:

1. Current active treatment with chemotherapy , radiation or surgery in the past 3 months or planned treatment during this study protocol period. Hormonal therapy is allowed.
2. Treatment with any neuropathic agent including taxane, platinum, vinca alkaloid, or bortezumab chemotherapy in the past 6 months.
3. Local infection at or near the acupuncture site. (Although acupuncture is a minimally invasive procedure, patients will be excluded if there is an indication of infection.)
4. Physical deformities that could interfere with accurate acupuncture point location.
5. Concurrent use of other alternative medicines such as herbal agents and high dose vitamins.
6. Known coagulopathy or taking heparin (including low molecular weight heparin) at full anti-coagulation doses (prophylaxis is allowed) or Coumadin at any dose. Patients on aspirin or non-steroidal anti-inflammatories or other antiplatelet medicines will be allowed to participate.
7. Platelets < 50 H K/UL in the past 30 days.
8. White blood cells (WBCs) < 3.0 K/UL or absolute neutrophil count (ANC) <1,500 K/UL) in the past 30 days.
9. Active central nervous system (CNS) disease. (The action for acupuncture may be associated with central nervous system activity, and patients with CNS pathology may respond differently to treatment than the general population.)
10. Cardiac pacemaker.
11. Mental incapacitation or significant emotional or psychological disorder that, in the opinion of the investigators, precludes study entry. (These patients may not be able to cooperate with this slightly invasive procedure or with the data collection process.)
12. Currently pregnant. (Certain acupuncture applications have been reported to stimulate uterine contractions.)
13. History of diabetic neuropathy or neuropathy related to HIV.
14. Previous acupuncture treatment for any indication within 30 days of enrollment.
15. Planned or actual changes in type of medications that could affect symptoms related to CIPN. New medications for the treatment of CIPN are not allowed during the study. Note: Subjects need to be on stable doses for 4 weeks.
16. Grade III lymphedema or lymphedema considered severe by the treating clinician.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-07-06 (Actual); Primary Completion 2016-05-10 (Actual); Study Completion 2016-05-10 (Actual)

PRIMARY OUTCOMES:
Score Changes in Neurotoxicity Scale | 4 weeks and 6 weeks
  Efficacy analysis used employing a paired t-test to estimate the mean changes in the score of the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group (FACT/GOG) Scale separately from baseline to after 12 treatments for each acupuncture schedule. 95% confidence intervals calculated for these estimates. T-test used to compare differences in scores (from baseline to after 12 treatments) between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Kay Garcia, DRPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org